CLINICAL TRIAL: NCT00361985
Title: Randomized, Prospective, Double-blind Trial of PPI vs Placebo in Prevention of Gastrojejunal Strictures After Laparoscopic Roux-en-Y Gastric Bypass for Morbid Obesity
Brief Title: Study of Proton Pump Inhibitors (PPI) to Prevent Strictures After Gastric Bypass Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Gregory Dakin, MD, Weill Cornell Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0511008254
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Anastomotic Stricture; Morbid Obesity
Keywords: Gastric bypass; Anastomotic stricture; Morbid obesity; Bariatric surgery; Omeprazole
MeSH Terms: conditions — Obesity, Morbid | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Nexium group
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 40mg once daily orally.
  Other Names: Nexium
Drug: Esomeprazole — Esomeprazole 40mg once daily orally
  Other Names: Nexium

SUMMARY:
The purpose of this study is to determine whether suppressing acid production by administration of daily proton pump inhibitors in the early post-operative period will reduce the gastrojejunal anastomosis stricture rate in patients undergoing laparoscopic gastric bypass surgery for morbid obesity.

DETAILED DESCRIPTION:
Laparoscopic Roux-en-Y gastric bypass (LYRGB) has been shown to be a safe and effective procedure for the treatment of morbid obesity. However, a common early complication of LYRGB is stricture at the gastrojejunal (GJ) anastomosis, occurring in 4% - 27% of patients, usually within the third post-operative month. This complication usually presents with progressive dysphagia leading to daily vomiting. Endoscopic balloon dilation is the treatment of choice for this complication, and multiple dilations are often required to provide complete resolution.

The etiology of GJ anastomotic strictures is unknown and is probably multi-factorial. Some investigators hypothesize that ischemia or non-ischemia-related excessive scar formation is the cause of stricture. The method of construction of the anastomosis as well seems to have an impact, as circular stapled anastomoses may have higher rates of stricture than linear staplers or completely hand-sewn anastomoses. The route of the Roux limb (antecolic vs retrocolic) does not appear to affect this complication.

Several investigators have demonstrated little acid production in the gastric bypass pouch. Despite this data, acid secretion has been hypothesized as a predominant factor in the development of GJ stricture. This hypothesis is supported in part by the frequent finding of ulcers at the site of stricture in up to 55% of patients. The purpose of this study is to determine whether suppressing acid production by administration of daily proton pump inhibitors in the early post-operative period will reduce GJ anastomosis stricture rate.

PLEASE NOTE: THIS STUDY DOES NOT PROVIDE SURGERY (APPROPRIATE INSURANCE COVERAGE IS REQUIRED).

ELIGIBILITY:
Inclusion Criteria:

* Any patient who satisfies the requirements of the Weill-Cornell Weight Loss Surgery program to undergo laparoscopic Roux-en-Y gastric bypass surgery as treatment for morbid obesity.

Exclusion Criteria:

* Patients with a history of ulcer disease, patients taking chronic acid suppression medicine, and patients taking NSAIDS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Gastrojejunal stricture | 6 months after surgery

SECONDARY OUTCOMES:
Gastrojejunal ulcer | 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gregory F. Dakin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell Unversity, New York, New York, United States